CLINICAL TRIAL: NCT04291976
Title: Back-to-back High-definition White Light Endoscopy Versus Single-pass High-definition White Light Endoscopy and Chromoendoscopy in IBD Surveillance
Brief Title: Back-to-back Endoscopy Versus Single-pass Endoscopy and Chromoendoscopy in IBD Surveillance
Acronym: HELIOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: UMC Utrecht (Other); Leiden University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109344
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Inflammatory Bowel Diseases; Colorectal Neoplasms
Keywords: IBD; Inflammatory Bowel Diseases; Colorectal Cancer; Surveillance; Dysplasia; Back-to-Back; Chromoendoscopy; White light
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a multicenter, non-blinded randomized trial with three parallel arms: back-to-back HDWLE, single-pass HDWLE and CE.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- back-to-back HDWLE (Experimental): Similar to single-pass HDWLE, with a second segmental inspection after the first examination in the same session. Equipment is similar to 1.
  Interventions: Procedure: Back-to-back high-definition white light endoscopy
- single-pass HDWLE (Active Comparator): Using HD white light, the entire colon is examined for dysplasia and other abnormalities after the caecum is reached. The colonoscope has a high-definition camera and processor. All images are displayed on a high definition monitor for optimal resolution.
  Interventions: Procedure: single-pass high-definition white light endoscopy
- Chromoendoscopy (Active Comparator): After introduction of the endoscope into the colon a dye (methylene blue or 0.3% indigo carmine) will be sprayed through a catheter positioned into the biopsy channel. Per segment, the entire colon is dyed, inspected, and lesions are removed. Equipment is similar to the other two arms.
  Interventions: Procedure: chromoendoscopy

INTERVENTIONS:
Procedure: Back-to-back high-definition white light endoscopy — Using HD white light, the entire colon is examined for dysplasia and other abnormalities after the caecum is reached, with a second segmental inspection after the first examination in the same session.The colonoscope has a high-definition camera and processor. All images are displayed on a high definition monitor for optimal resolution.
  Arms: back-to-back HDWLE
Procedure: single-pass high-definition white light endoscopy — Using HD white light, the entire colon is examined for dysplasia and other abnormalities after the caecum is reached. The colonoscope has a high-definition camera and processor. All images are displayed on a high definition monitor for optimal resolution.
  Arms: single-pass HDWLE
Procedure: chromoendoscopy — After introduction of the endoscope into the colon a dye (methylene blue or indigo carmine) will be sprayed through a catheter positioned into the biopsy channel. Per segment, the entire colon is dyed, inspected, and lesions are removed. Equipment is similar to the other two interventions.
  Arms: Chromoendoscopy

SUMMARY:
The current international guidelines for CRC surveillance in IBD recommend as first choice the use of chromoendoscopy, and as an alternative high-definition white light endoscopy (HDWLE) for optimal dysplasia detection, based on data from clinical trials. However, data on the superiority of CE over HDWLE are not consistent in literature. The investigators hypothesize that the better performance of CE in some clinical trials is the result of the associated longer procedural time and the fact that every colon segment is examined twice. Currently, no studies have been published evaluating the dysplastic yield of back-to back HDWLE compared to HDWLE with a single pass or CE in patients with IBD. In the present study, the investigators aim to compare the yield of dysplasia/CRC between 1) regular HDWLE, 2) HDWLE back-to-back, and 3) CE.

DETAILED DESCRIPTION:
The investigators assume based on previous research a yield of 12% using high-definition white light endoscopy and 24% using either chromoendoscopy or high-definition white light endoscopy with a second examination (Imperatore et al 2019). To show non-inferiority of back-to-back HDWLE compared to CE, with a non-inferiority margin of 10% (power 80% and alpha 5%,) a total of 226 patients per group is required.

To demonstrate a superiority of back-to-back HDWLE compared to a regular HDWLE, with a 1:2 allocation ratio of single-pass vs back-to-back , 113 and 226 patients per group are needed to achieve 80% power with an alpha of 5%. Therefore, the investigators will include 226 patients in group back-to-back HDWLE, 226 in group CE, and 113 patients in group regular HDWLE. This amounts to a total of 560 patients. To account for any screen-failures The investigators will include at most 5% (of 560) additional patients until 80% power is reached.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients with inflammatory bowel disease, an estimated involvement of at least 30% of the colonic surface and a disease duration of at least 8 years (or any disease duration in case of concomitant primary sclerosing cholangitis).
* Previous assessable surveillance endoscopy > 1 year
* Age > 18 years

Exclusion Criteria:

* Active colitis > 20 cm and/or inflammation resulting in an insufficient surveillance procedure according to the endoscopist.
* Allergy or intolerance to methylene blue
* Insufficient bowel cleansing (BBPS <6)
* Refusing or incapable to agree with informed consent
* Pregnant women
* > 50 % of the colon surgically removed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
detection rate of neoplasia for each technique | During endoscopy

SECONDARY OUTCOMES:
Number of all lesions for each technique | During endoscopy
Number of dysplastic lesions for each technique | After each endoscopy, within one month after the procedure.
Kudo classification for each lesion | During endoscopy when a lesion is detected
Duration | During endoscopy
  Total endoscopic procedure time and endoscopic procedure time during withdrawal for each technique.
Number of targeted biopsies taken in the different groups. | During endoscopy
Percentage of non-interpretable/assessable endoscopies | During endoscopy
  e.g. insufficient preparation, inflammation
Location of the lesion | During endoscopy
Size of the lesion in mm | During endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hoentjen, MD PhD, Principal Investigator — Radboud University Medical Center; Bas Oldenburg, MD PhD, Principal Investigator — UMC Utrecht
Locations (4):
- Netherlands (4):
  - Radboudumc, Nijmegen, Gelderland
  - Utrecht University Medical Center, Utrecht, Gelderland
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
  - Leiden University Medical Center, Leiden, South Holland

IPD SHARING:
Plan to Share IPD: No